CLINICAL TRIAL: NCT02191631
Title: Internet-delivered Cognitive Behavior Therapy for Adolescents With Obsessive-Compulsive Disorder: A Randomized Controlled Study
Brief Title: Internet-delivered CBT for Adolescents With OCD: A Randomized Controlled Study
Acronym: BiPOCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Serlachius, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiPOCD RCT
Record Dates: First submitted 2014-07-03; First posted 2014-07-16 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; adolescents; pediatric; internet; online; CBT
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-delivered CBT (Experimental): Participants will receive 12 weeks of internet-delivered cognitive behavior therapy with psychologist support.
  Interventions: Behavioral: Internet-delivered Cognitive Behavior Therapy
- Wait list (No Intervention): Participants will receive no treatment for 12 weeks. After that period participants will receive Internet-delivered Cognitive Behavior Therapy.

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavior Therapy — The treatment consists of standard cognitive behavior therapy for obsessive-compulsive disorder and is delivered via an internet plattform and regular therapist contact several times per week via email and telephone. The treatment is 12 weeks.
  Arms: Internet-delivered CBT

SUMMARY:
The effect of Internet-delivered Cognitive Behavior Therapy (ICBT) on adolescents (12 to 17 years) with Obsessive-Compulsive Disorder is studied. Participants are randomized to either ICBT or a no-treatment condition. We expect ICBT to be superior over the no-treatment condition.

DETAILED DESCRIPTION:
The primary objective of this study is to test the efficacy of Internet-delivered cognitive behavior therapy (ICBT) for adolescents (12 - 17 years) with OCD. We aim to conduct a randomized controlled study with N = 66 participants. Participants will be randomly assigned to ICBT or a wait list condition, either lasting 12 weeks. The primary outcome measure is the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS). Study participants will be followed up 3 and 12 months after treatment. ICBT is expected to yield significantly better symptom reduction than the wait list condition.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of OCD as defined by DSM-5
* a total score of ≥ 16 on the Children's Yale-Brown Obsessive-Compulsive Scale, CY-BOCS
* age between 12 and 17 years
* ability to read and write Swedish
* daily access to the internet
* a parent that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* diagnosed autism spectrum disorder, psychosis or bipolar disorder, severe eating disorder
* suicidal ideation
* ongoing substance dependence
* subject not able to read or understand the basics of the ICBT material
* completed CBT for OCD within last 12 months (defined as at least 5 sessions of CBT including exposure and response prevention)
* ongoing psychological treatment for OCD or another anxiety disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive Compulsive Scale, CY-BOCS | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Change from Baseline of obsessions and compulsions after 12 weeks and at 3- and 12 months after treatment

SECONDARY OUTCOMES:
Clinical Global Impression - Severity, CGI-S | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Clinical Global Impression - Improvement, CGI-I | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Parent Adherence EX/RP Scale, PEAS | Baseline, 6 and 12 weeks after treatment starts
Children's Obsessional Compulsive Inventory Revised, (CHOCI-R, Shafran et al., 2003) | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Education, Work and Social Adjustment Scale - child and parent version (EWSAS) | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Spence Child Anxiety Scale - Child and Parent version (SCAS-C/P, Spence, 1998 | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Child Depression Inventory - Short version (CDI-S, Kovacs, 1985) | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Family Accommodation Scale, Parent-Report (FAS-PR, Flessner et al., 2009) | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
Technology acceptance scale | Baseline, 6 and 12 weeks after treatment starts,
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness - Child version (TiC-P) | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
EQ-5D - quality of life | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended

OTHER OUTCOMES:
Measurement of homework adherence | Baseline, daily measurements until 12 weeks after baseline
Number of Participants with Adverse Events | 12 weeks after baseline
DNA samples (from blood and/or saliva) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lenhard F, Ssegonja R, Andersson E, Feldman I, Ruck C, Mataix-Cols D, Serlachius E. Cost-effectiveness of therapist-guided internet-delivered cognitive behaviour therapy for paediatric obsessive-compulsive disorder: results from a randomised controlled trial. BMJ Open. 2017 May 17;7(5):e015246. doi: 10.1136/bmjopen-2016-015246. PMID 28515196
- [Derived] Lenhard F, Andersson E, Mataix-Cols D, Ruck C, Vigerland S, Hogstrom J, Hillborg M, Brander G, Ljungstrom M, Ljotsson B, Serlachius E. Therapist-Guided, Internet-Delivered Cognitive-Behavioral Therapy for Adolescents With Obsessive-Compulsive Disorder: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2017 Jan;56(1):10-19.e2. doi: 10.1016/j.jaac.2016.09.515. Epub 2016 Oct 25. PMID 27993223